CLINICAL TRIAL: NCT05597215
Title: Two Bed SPECT/CT Versus Planar Bone Scintigraphy in Detection of Osseous Metastases in Patients With Genitourinary Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maram Mostafa Shafeek, Principal investigator, Assiut University
Other Study IDs: Tc-99m MDP bone scintigraphy
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Bone Metastases; Urogenital Cancer
Keywords: Bone scintigraphy
MeSH Terms: conditions — Urogenital Neoplasms | interventions — Technetium Tc 99m Medronate; Gamma Cameras

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Tc-99m MDP and gamma camera — Injection of radioactive element (Tc-99m MDP) then imaging with gamma camera and low dose CT (SPECT/CT)

SUMMARY:
The study aims to compare the diagnostic performance of planar bone scan and two bed SPECT/CT in detection of bone metastases in patients with urogenital cancer.

DETAILED DESCRIPTION:
Genitourinary malignancies represent a heterogeneous group of diseases linked by anatomical and physiological function. Renal cell carcinoma (RCC); urothelial carcinoma of the bladder, ureter, and renal pelvis, and prostate adenocarcinoma (PC) are the most commonly encountered histological subtypes within this group. Planar bone scintigraphy (PBS) with di-phosphonate compounds is widely used, cost-effective and sensitive imaging modality for detecting osseous metastases especially in prostate cancer. However, it suffers from low specificity as well as low sensitivity in purely osteolytic lesions. Single-photon emission computed tomography (SPECT) is a three-dimensional acquisition method that has demonstrated greater sensitivity and specificity compared to planar images, especially for detecting vertebral metastases. The introduction of SPECT/CT images improves the lesion-to-background ratio, allows anatomic lesion localization, removes the superimposition of anatomical structures, such as urinary bladder activity, and provides anatomical data, thereby increasing the sensitivity, specificity and positive predictive value of bone scan. As the technology advances, current SPECT/CT machines have become capable of sequentially covering, and accurately merging, more than one field of view (FOV) in a reasonable time. In this study, we aim to compare the diagnostic performance of two-bed SPECT/CT images and planar bone scintigraphy in detection of bone metastases in genitourinary malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with urogenital cancer referred for bone scan.

Exclusion Criteria:

* Patients with claustrophobia.
* Patients refuse to do the scan.
* Patients with relative or absolute contraindications to do the scan (eg. pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with known genitourinary cancer who are referred for bone scan as a part of metastatic workup.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of diagnostic performance indices between two-bed SPECT/CT images and planar bone scans. | through study completion, an average of 2 years
  Analysis and comparison of diagnostic performance indices between two-bed SPECT/CT images and planar bone scans for the detection of osseous metastases in genitourinary malignancies.

SECONDARY OUTCOMES:
Identification of patients' subgroups who might be best assessed upfront by two-bed SPECT/CT. | through study completion, an average of 2 years
Identification of anatomical site which may be best assessed by SPECT/CT. | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samir S Mohamed, Professor, Study Chair — Assiut University; HebatAllah A Askar, Lecturer, Study Director — Assiut University; Rehab M Helmy, Lecturer, Study Director — Assiut University; Maram M Shafeek, Resident, Principal Investigator — Assiut University

REFERENCES:
- [Background] Zarrabi K, Paroya A, Wu S. Emerging therapeutic agents for genitourinary cancers. J Hematol Oncol. 2019 Sep 4;12(1):89. doi: 10.1186/s13045-019-0780-z. PMID 31484560
- [Background] Costa WH, Jabboure G Netto, Cunha IW. Urological cancer related to familial syndromes. Int Braz J Urol. 2017 Mar-Apr;43(2):192-201. doi: 10.1590/S1677-5538.IBJU.2016.0125. PMID 27819754
- [Background] Van den Wyngaert T, Strobel K, Kampen WU, Kuwert T, van der Bruggen W, Mohan HK, Gnanasegaran G, Delgado-Bolton R, Weber WA, Beheshti M, Langsteger W, Giammarile F, Mottaghy FM, Paycha F; EANM Bone & Joint Committee and the Oncology Committee. The EANM practice guidelines for bone scintigraphy. Eur J Nucl Med Mol Imaging. 2016 Aug;43(9):1723-38. doi: 10.1007/s00259-016-3415-4. Epub 2016 Jun 4. PMID 27262701
- [Background] Rager O, Nkoulou R, Exquis N, Garibotto V, Tabouret-Viaud C, Zaidi H, Amzalag G, Lee-Felker SA, Zilli T, Ratib O. Whole-Body SPECT/CT versus Planar Bone Scan with Targeted SPECT/CT for Metastatic Workup. Biomed Res Int. 2017;2017:7039406. doi: 10.1155/2017/7039406. Epub 2017 Jul 24. PMID 28812019
- [Background] Umer M, Mohib Y, Atif M, Nazim M. Skeletal metastasis in renal cell carcinoma: A review. Ann Med Surg (Lond). 2018 Jan 31;27:9-16. doi: 10.1016/j.amsu.2018.01.002. eCollection 2018 Mar. PMID 29511536
- [Background] Shen G, Deng H, Hu S, Jia Z. Comparison of choline-PET/CT, MRI, SPECT, and bone scintigraphy in the diagnosis of bone metastases in patients with prostate cancer: a meta-analysis. Skeletal Radiol. 2014 Nov;43(11):1503-13. doi: 10.1007/s00256-014-1903-9. Epub 2014 May 20. PMID 24841276
- [Background] de Leiris N, Leenhardt J, Boussat B, Montemagno C, Seiller A, Phan Sy O, Roux J, Laramas M, Verry C, Iriart C, Fiard G, Long JA, Descotes JL, Vuillez JP, Riou L, Djaileb L. Does whole-body bone SPECT/CT provide additional diagnostic information over [18F]-FCH PET/CT for the detection of bone metastases in the setting of prostate cancer biochemical recurrence? Cancer Imaging. 2020 Aug 12;20(1):58. doi: 10.1186/s40644-020-00333-y. PMID 32787923
- [Background] Zacho HD, Manresa JAB, Aleksyniene R, Ejlersen JA, Fledelius J, Bertelsen H, Petersen LJ. Three-minute SPECT/CT is sufficient for the assessment of bone metastasis as add-on to planar bone scintigraphy: prospective head-to-head comparison to 11-min SPECT/CT. EJNMMI Res. 2017 Dec;7(1):1. doi: 10.1186/s13550-016-0252-1. Epub 2017 Jan 5. PMID 28058659